CLINICAL TRIAL: NCT02861755
Title: Online Positive Emotion Skills Intervention for Symptoms of Depression (MARIGOLD)
Brief Title: Online Positive Emotion Skills Intervention for Symptoms of Depression
Acronym: MARIGOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of California, San Francisco (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Judith Moskowitz, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00092507; R34MH101265-02 (NIH)
Record Dates: First submitted 2016-06-13; First posted 2016-08-10 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Depression; Psychological Stress; Affect
Keywords: Depression; Depressive Disorder; Psychological Stress; Behavioral Symptoms; Mental Disorders; Mood Disorders
MeSH Terms: conditions — Depression; Stress, Psychological; Depressive Disorder; Behavioral Symptoms; Mental Disorders; Mood Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental): The MARIGOLD positive emotions course plus a blend of enhancements to include: 5-minutes of weekly facilitator contact, online discussion board, or gamification through virtual flower badges.
  Interventions: Behavioral: Positive Affect Skills Training
- Arm 2 (Experimental): Emotion reporting control condition. Reporting daily emotions for the same duration of the online emotions course.
  Interventions: Behavioral: 5-week Emotion Reporting

INTERVENTIONS:
Behavioral: Positive Affect Skills Training — Blend of enhancements may include: 5-minutes of facilitator contact, an online discussion board, or gamification via virtual flower badges.
  Arms: Arm 1
Behavioral: 5-week Emotion Reporting
  Arms: Arm 2

SUMMARY:
Major depressive disorder affects over 120 million people worldwide. Only 50% of Americans with depression receive adequate treatment, and one-third of those receiving treatment do not benefit. In this pilot project investigators will bring together two approaches that have the promise to reach large numbers of depression sufferers: a skills-based intervention for increasing positive affect and experiences in depressed individuals, delivered in an inexpensive self-paced mobile format. The study will make use of smartphone technology to improve conventional outcome measurement via in-the-moment emotion sampling and mobile assessment of heart rate variability, a predictor of cardiac health that may mediate some of the health effects of depression. The aims are: 1) Retool the existing web-based positive emotion intervention for use on smartphones, with innovative exercises that help participants bring the skills they are learning into real-life situations; 2) Perform a small feasibility trial of the mobile intervention on individuals with clinical depression recruited online 3) Eventually incorporate feedback from the small feasibility trial to improve the online intervention and conduct a full randomized trial on a larger scale

ELIGIBILITY:
Inclusion Criteria:

* Daily internet access
* Cell phone ownership
* Score of 5 or higher on PHQ-8 scale
* Lives in US or Canada
* Speaks and reads English, able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change in Retention Over Time (average of 4.5 months through study completion) | From the start of the 5-week online intervention (Weeks 1-5), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18). Data collected for the duration of the entire study.
  Determine the percentage of participants providing data at each stage of the study from baseline to study completion (average of 4.5 months). This includes capturing dropout rates and reasons for dropping out, where possible; Retention will also include analyzing any qualitative comments/feedback on the lessons and home practice exercises in order to gauge what participants like and don't like, and what is feasible for future iterations of this study to maximize retention.
Change in Depression symptoms (PHQ-8 questionnaire) Over Time (4.5 months through study completion) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  8-items; responses range from 0 "not at all" to 3 "almost every day"
Change in Depression symptoms (CES-D questionnaire) Over Time | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  20-items; responses range from 1 "rarely or none of the time (less than 1 day)" to 3 "occasionally or a moderate amount of the time (3-4 days)"

SECONDARY OUTCOMES:
Change in Stress: Perceived Stress Scale (PSS questionnaire) Over Time | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  10-items; responses range from 1 "never" to 5 "very often"
Change in Positive and Negative Affect (DES questionnaire) Over Time ("past week") | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  26-items; responses range from 1 "not at all" to 9 "all the time"; framed as "Over the PAST week, how much have you felt each of these emotions?"
Change in Mindfulness Over Time: Five Facet Mindfulness Questionnaire (FFMQ) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  7-items; responses range from 1 "never or rarely true" to 5 "very often or always true"
Change in Prioritizing Positivity Over Time (Prioritizing Positivity Scale) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  6-items; responses range from 1 "disagree strongly" to 9 "agree strongly"
Skills Use Questionnaire (measuring change in application/use of positive affect skills over 4.5 months) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  10-items; responses range from 1 "definitely false" to 5 "definitely true"
Change in Brief Resilience Scale (BRS) over time (4.5 months of participation in the study) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  6-items of self-reported resilience; responses range from 1 "strongly disagree" to 5 "strongly agree"
Change in Depression Self Stigma Scale (DSSS) over time (4.5 months of participation in the study) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  32-item scale to measure self stigma of depression; responses range from 1 "completely disagree" to 7 "completely agree"
Change in Meaning and Purpose Scale over time (4.5 months of participation in the study) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  8-item scale with 5 response options ranging from "strongly disagree" to "strongly agree"
Change in Positive Affect and Well-Being Short Form from the Neuro-QOL Item Bank | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  9-item scale measuring positive affect and well-being with 5 response options: "never" "rarely" "sometimes" "often" "always"
Change in General Behavior Inventory (GBI) Scale | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  7-item instrument assessing for symptoms of mania with 7 response options: 0 "Never or hardly ever," 1 "Sometimes," 2 "Often," 3 "Very Often," 7 "Don't Know," 8 "Refuse to Answer," 9 "Not applicable." The 7 items include questions such as: "Have there been times lasting several days or more when you felt you must have lots of excitement, and you actually did a lot of new or different things?"
Change in Behavioral Activation for Depression Scale (BADS) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  9-item instrument that measures the impact of behavioral activation on depressive symptoms. Response items range from 0 to 6, from "Not at all" to "Completely." Statements include: "I was an active person and accomplished the goals I set out to do" and "I did things that were enjoyable."
Change in Stress Management Self-Efficacy (SMSE) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  4-item instrument that measures the impact of stress on depressive symptoms. Response scale ranges from 1 "strongly agree" to 4 "strongly disagree." Items include: 1) I believe I have the ability to cope with the demands of my life 2) I know when I'm starting to experience too much stress 3) I know how to cope with stress when it comes and 4) I am usually able to successfully deal with my stress levels.
Expectancy Credibility Scale | Administered once at the initial questionnaire prior to Week 1 of the intervention.
  6-item instrument that measures how expectancy and credibility might influence participants' responses. Responses range from 1 "Not at all" to 9 "Very." Statements include: "At this point, how logical does this course seem to you?" or "At this point, how much do you really feel that the course will help you to improve your functioning?"
Change in Self Compassion Scale (SCS) Short-Form | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  12-item instrument assesses levels of self-compassion. Response items range from 1 "Almost never" to 5 "Almost always." Statements include: "I try to see my failings as part of the human condition" and "When something painful happens I try to take a balanced view of the situation."
Change in Self-Stigma Depression Scale (SSDS) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  16-item instrument that assesses levels of self-stigma surrounding depressive symptoms. This measure will be used to replace the DSSS from the pilot phase of the study.

OTHER OUTCOMES:
Change in Life Satisfaction Scale | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  ratings of life, job, relationship on a 9-point scale, from 1 "not satisfied" to 9 "satisfied"
Change in Burnout Scale | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  rating health and sleep quality on a 9-point scale from 1 "poor" to 9 "excellent"
Change in Importance of Happiness (1-item measure) | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  1 item measure on a 9-point scale ranging from 1 "not very important" to 9 "very important"
Change in Personality Scale | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  self-rated personality for dependability/discipline and disorganization/carelessness on a 9-point scale from 1 "strongly disagree" to 9 "strongly agree."
Change in Daily Inventory of Stressful Events (DISE) Self-Assessment over 5 weeks (daily) | Starts at the onset of the 5-week intervention (Week 1) and continues throughout the 5 weeks on a daily basis (through Week 5)
  7-items measuring stressful events with 5 response items ranging from 0 "didn't happen" to 4 "very stressful"
Change in Differential Emotions Scale (DES) over 5 weeks (daily) | Starts at the onset of the 5-week intervention (Week 1) and continues throughout the 5 weeks on a daily basis (through Week 5)
  26-items; responses range from 1 "not at all" to 9 "all the time"; framed as "Over the PAST day, how much have you felt each of these emotions?"
Change in self-reported mental health status | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  6 self-report questions asking about depression diagnosis, medication, therapies, treatment. For example, "Have you ever taken medication for anxiety, worry, or stress?" with options such as "I'm currently taking medication" "In the past, but not now" and "No."
Change in Happiness Inducing Behavior (HIB) Scale | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  38-items assessing how often repondents have completed happiness inducing behaviors. Adapted scale and 7 response options range from "Not at all" to "Multiple Times a Day"
Change in Situational Motivation Scale (SIMS) | Post-intervention (Week 6), 1 month followup (Week 10), and 3 month followup (Week 18) only
  16-items assessing what motivates a respondent to use the MARIGOLD skills with 7 response options ranging from 1 "Not at all" to 7 "Exactly"
Technology Survey | Administered only at baseline (Week 1) and post-intervention (Week 6).
  6-items administered at baseline to assess level of technology use, modes of use, and frequency of use. 1-item technology question at post-intervention asking which device participants used the most for MARIGOLD.
Change in Pain | From the start of the 5-week online intervention (Week 1), post-intervention (Week 6), 1 month followup (Week 10), 3 month followup (Week 18).
  Single-Item pain measure assessed at each timepoint to measure change in pain level. Asks about the average level of pain over the past week on a scale of 0 to 10, with 0 being "No pain" and 10 being "Pain as bad as you can imagine."

CONTACTS AND LOCATIONS:
Overall Officials: Judith T Moskowitz, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, MSS Dept, Chicago, Illinois, United States

REFERENCES:
- [Background] Moskowitz JT, Hult JR, Duncan LG, Cohn MA, Maurer S, Bussolari C, Acree M. A positive affect intervention for people experiencing health-related stress: development and non-randomized pilot test. J Health Psychol. 2012 Jul;17(5):676-92. doi: 10.1177/1359105311425275. Epub 2011 Oct 21. PMID 22021272
- [Derived] Moskowitz JT, Jackson K, Freedman ME, Grote VE, Kwok I, Schuette SA, Cheung EO, Addington EL. Positive Psychological Intervention Effects on Depression: Positive Emotion Does Not Mediate Intervention Impact in a Sample with Elevated Depressive Symptoms. Affect Sci. 2022 Oct 6;4(1):163-173. doi: 10.1007/s42761-022-00140-7. eCollection 2023 Mar. PMID 37070017
- [Derived] Moskowitz JT, Addington EL, Shiu E, Bassett SM, Schuette S, Kwok I, Freedman ME, Leykin Y, Saslow LR, Cohn MA, Cheung EO. Facilitator Contact, Discussion Boards, and Virtual Badges as Adherence Enhancements to a Web-Based, Self-guided, Positive Psychological Intervention for Depression: Randomized Controlled Trial. J Med Internet Res. 2021 Sep 22;23(9):e25922. doi: 10.2196/25922. PMID 34550076
- [Derived] Cheung EO, Addington EL, Bassett SM, Schuette SA, Shiu EW, Cohn MA, Leykin Y, Saslow LR, Moskowitz JT. A Self-Paced, Web-Based, Positive Emotion Skills Intervention for Reducing Symptoms of Depression: Protocol for Development and Pilot Testing of MARIGOLD. JMIR Res Protoc. 2018 Jun 5;7(6):e10494. doi: 10.2196/10494. PMID 29871853